CLINICAL TRIAL: NCT00025675
Title: ZD1839 FOR Treatment Of Recurrent Or Progressive Malignant Astrocytoma Or Glioblastoma And Recurrent Or Progressive Meningioma: A Phase II Study With A Phase I Component For Patients Receiving EIAEDs
Brief Title: Gefitinib in Treating Patients With Recurrent or Progressive CNS Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NABTC-0001 CDR0000068984; U01CA062399 (NIH); ABTC-0001; NABTC-0001
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult meningioma; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult pilocytic astrocytoma; adult subependymoma; adult mixed glioma; adult meningeal hemangiopericytoma; adult grade III meningioma; adult giant cell glioblastoma; adult gliosarcoma; adult grade I meningioma; adult grade II meningioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Meningioma; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma, Subependymal; Glioma; Gliosarcoma | interventions — Gefitinib

ARMS (2):
- p450 (Active Comparator): p450 inhibitor
  Interventions: Drug: gefitinib
- nonp450 (Active Comparator): not on p450 inhibitor
  Interventions: Drug: gefitinib

INTERVENTIONS:
Drug: gefitinib

SUMMARY:
RATIONALE: Biological therapies such as gefitinib may interfere with the growth of tumor cells and slow the growth of CNS tumors.

PURPOSE: Phase II trial to study the effectiveness of gefitinib in treating patients who have recurrent or progressive CNS tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of gefitinib in patients with recurrent or progressive supratentorial malignant gliomas or brain or spinal meningiomas receiving enzyme-inducing antiepileptic drugs (EIAEDs). (Phase I of the study closed to accrual as of 09/19/2003).
* Determine the toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in patients receiving EIAEDs.
* Determine the efficacy of this drug in terms of 6-month progression-free survival of these patients.
* Determine the safety profile of the phase II dose of this drug in these patients.

OUTLINE: This is a multicenter, dose-escalation study. Patients are stratified according to concurrent enzyme-inducing antiepileptic drugs (EIAEDs) (yes vs no) and disease type (for phase II only) (benign meningioma vs malignant meningioma vs hemangiopericytoma vs glioblastoma vs other anaplastic glioma). (Phase I closed to accrual as of 09/19/2003).

Patients receive oral gefitinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients (who are receiving EIAEDs) receive escalating doses of gefitinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 2 weeks.

PROJECTED ACCRUAL: A minimum of 30 patients will be accrued for the phase I portion of this study within 10 months . (Phase I closed to accrual as of 09/19/2003). A total of 48 patients will be accrued for the phase II portion of this study within 6-8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Histologically confirmed supratentorial malignant primary glioma

    * Glioblastoma multiforme
    * Anaplastic astrocytoma
    * Anaplastic oligodendroglioma
    * Anaplastic mixed oligoastrocytoma
    * Malignant astrocytoma not otherwise specified
  * Histologically confirmed or radiographically defined recurrent or progressive brain or spinal meningioma, including base of skull or cavernous sinus meningiomas

    * Benign, malignant, or atypical
    * May include neurofibromatosis type I or II
    * Hemangiopericytoma allowed
* Recurrent or progressive disease by MRI or CT scan

  * Evidence of true progressive disease by PET or thallium scan, MR spectroscopy, or surgical documentation required if patient received prior interstitial brachytherapy or stereotactic radiosurgery (to the target lesion for meningioma and hemangiopericytoma)
  * Steroid dosage must be stable for at least 5 days prior to scan
* No limitations on the number of prior surgeries, radiotherapy or chemotherapy regimens, or radiosurgery treatments for patients with meningioma or hemangiopericytoma and may include standard external beam radiotherapy, interstitial brachytherapy, or gamma-knife radiosurgery in any combination
* Patients with glioma must have failed prior radiotherapy
* Original histology of low-grade glioma allowed if subsequent confirmation of malignant glioma is made at time of recurrence
* Phase I (closed to accrual as of 09/19/2003):

  * Prior treatment for no more than 3 prior relapses in patients with glioma
* Phase II:

  * Measurable disease after prior surgical resection of recurrent or progressive disease
  * Prior treatment for no more than 2 prior relapses in patients with glioma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 8 weeks

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 120,000/mm^3
* Hemoglobin at least 10 g/dL (transfusion allowed)

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT less than 1.5 times ULN

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No significant cardiac risk factors within the past 6 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No gastrointestinal risk factors (e.g., active ulcerative colitis) within the past 6 months
* No active infection
* No concurrent disease that would obscure toxicity or dangerously alter drug metabolism
* No other significant medical illness that would preclude study
* No other malignancy within the past 3 years except non-melanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior interferon or thalidomide
* No concurrent filgrastim (G-CSF)

Chemotherapy:

* See Disease Characteristics
* At least 2 weeks since prior vincristine
* At least 6 weeks since prior nitrosoureas
* At least 3 weeks since prior procarbazine

Endocrine therapy:

* At least 1 week since prior tamoxifen

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics
* At least 7 days since prior surgery for recurrent or progressive tumor and recovered

Other:

* Recovered from prior therapy
* No prior gefitinib or other epidermal growth factor receptor inhibitor
* At least 1 week since prior isotretinoin
* At least 1 week since other prior noncytotoxic agents (except radiosensitizers)
* At least 4 weeks since prior investigational agents
* Concurrent low-molecular weight heparin or warfarin for deep vein thrombosis or pulmonary embolism allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2001-10-09 (Actual); Primary Completion 2006-07-05 (Actual); Study Completion 2010-01-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank S. Lieberman, MD, Study Chair — University of Pittsburgh
Locations (12):
- United States (12):
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Neuro-Oncology Branch, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Background] Norden AD, Raizer JJ, Abrey LE, Lamborn KR, Lassman AB, Chang SM, Yung WK, Gilbert MR, Fine HA, Mehta M, Deangelis LM, Cloughesy TF, Robins HI, Aldape K, Dancey J, Prados MD, Lieberman F, Wen PY. Phase II trials of erlotinib or gefitinib in patients with recurrent meningioma. J Neurooncol. 2010 Jan;96(2):211-7. doi: 10.1007/s11060-009-9948-7. Epub 2009 Jun 28. PMID 19562255
- [Background] Lassman AB, Rossi MR, Raizer JJ, Abrey LE, Lieberman FS, Grefe CN, Lamborn K, Pao W, Shih AH, Kuhn JG, Wilson R, Nowak NJ, Cowell JK, DeAngelis LM, Wen P, Gilbert MR, Chang S, Yung WA, Prados M, Holland EC. Molecular study of malignant gliomas treated with epidermal growth factor receptor inhibitors: tissue analysis from North American Brain Tumor Consortium Trials 01-03 and 00-01. Clin Cancer Res. 2005 Nov 1;11(21):7841-50. doi: 10.1158/1078-0432.CCR-05-0421. PMID 16278407